CLINICAL TRIAL: NCT05882240
Title: Evaluation of the Correct Performance and Knowledge About the Passive Leg Raise Test to Detect a Volume Reagibility in Critical Care Patients.
Brief Title: Performance of PLR as Predicting Preload Responsiveness
Acronym: PLR
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: JohannesGUVT
Record Dates: First submitted 2023-05-11; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Stroke Volume
Keywords: passive leg raise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: choice of initial position — current practice of correct application and interpretation of the PLR in critical care patients
  Other Names: Measurement of effect size

SUMMARY:
We aimed to establish current practice of correct application and interpretation of the PLR in critical care patients.

DETAILED DESCRIPTION:
The points of concern for PLR include the following: the indication and contraindication of PLR; the choice of initial position: starting from a semi-recumbent position or supine position for PLR; how to interpret and apply the changes of CO, blood pressure, and central venous pressure (CVP) to identify fluid response during PLR; and how to identify spontaneous variation and sympathetic stimulation during PLR.

ELIGIBILITY:
Inclusion Criteria:

* All Critical care physicians of different medical disciplines

Exclusion Criteria:

* not completely responses

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All Critical care physicians
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
We aimed to establish current practice of correct application and interpretation of the PLR in critical care patients | through study completion, an average of Measurement in 5 Minutes
  Application and Interpretation of correct effect size

SECONDARY OUTCOMES:
Profession | < 10 Minutes
  Profession of the respondents
Measurement of cardiac output | < 10 Minutes
  correct response of stroke volume

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, Principal Investigator — University Medical Centre
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No